CLINICAL TRIAL: NCT05618184
Title: Health-related Quality of Life Among Hungarian Women with Urinary Incontinence
Brief Title: Quality of Life Among Hungarian Women with Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Other Study IDs: BMEÜ/379-3/2022/EKU-2
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Urinary Incontinence
Keywords: Quality of life
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to assess the prevalence of urinary incontinence among Hungarian women. In addition to that, we aim evaluate the health related quality of life among Hungarian women with urinary incontinence and to culturally adapt the following questionnaires for the Hungarian population: Incontinence Impact Questionnaire - Short Form (IIQ-7) and King's Health Questionnaire (KHQ).

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Age 18 and above
* Providing consent to participate
* Ability to read and write Hungarian

Exclusion Criteria:

* Respondents who are unable to complete the online survey due to illiteracy
* Man

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years or older who are able to read and write Hungarian.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
International Consultation of Incontinence Questionnaire - Short Form | Baseline
  The International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF) will be used to gather information about the symptoms of urinary incontinence. It contains six questions. The total score can range from 0 to 21, with higher scores suggesting more severe symptoms.
King's Health Questionnaire | Baseline
  The King's Health Questionnaire (KHQ) will be used to measure the impact of urinary incontinence on the subject's health related quality of life. It assesses quality of life in nine different domains of life. Each domain is scored separately ranging from 0 (best) to 100 (worst).
Incontinence Impact Questionnaire short form | Baseline
  The Incontinence Impact Questionnaire short form (IIQ-7) will be also used to measure the impact of urinary incontinence on the subject's health related quality of life. It is comprised of seven questions. The total score ranges from 0 to 21, with higher scores indicating more severe symptoms and worse quality of life.

SECONDARY OUTCOMES:
Short-Form-36 | Baseline
  The Short-Form-36 (SF-36) will be used to measure the generic health-related quality of life of participants. It consists of 35 individual questions and it is divided into eight domains of health.
  The total score ranges from 0 (worst health state) to 100 (best health state).

CONTACTS AND LOCATIONS:
Overall Officials: Márta Hock, Habilitation, Principal Investigator — University of Pecs
Locations (1):
- University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: Undecided